CLINICAL TRIAL: NCT00791011
Title: A Phase 1b Study to Evaluate the Safety and Tolerability of AMG 655 in Combination With Bortezomib or Vorinostat in Subjects With Relapsed or Refractory Lymphoma
Brief Title: Phase 1b Lymphoma Study of AMG 655 in Combination With Bortezomib or Vorinostat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20060340
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Hodgkin's Lymphoma; Low Grade Lymphoma; Lymphoma; Mantle Cell Lymphoma; Non-Hodgkin's Lymphoma; Diffuse Large Cell Lymphoma
Keywords: Lymphoma; AMG 655; Trail receptor; Apoptosis; Vorinostat; Bortezomib; SAHA; Velcade
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — conatumumab; Vorinostat; Bortezomib

ARMS (7):
- Cohort 4 (Experimental): AMG 655 (intermediate dose) with Vorinostat
  Interventions: Drug: AMG 655; Other: Vorinostat
- Cohort 1 (Experimental): AMG 655 (low dose) with Bortezomib
  Interventions: Drug: AMG 655; Other: Bortezomib
- Cohort 2 (Experimental): AMG 655 (low dose) with vorinostat
  Interventions: Drug: AMG 655; Other: Vorinostat
- Cohort 5 (Experimental): AMG 655 (high dose) with Bortezomib
  Interventions: Drug: AMG 655; Other: Bortezomib
- Cohort 6 (Experimental): AMG 655 (high dose) with Vorinostat
  Interventions: Drug: AMG 655; Other: Vorinostat
- Cohort 7 (Experimental): Part 2 - Mantle Cell Lymphoma subjects only: AMG 655 at dose TBD with Bortezomib
  Interventions: Drug: AMG 655; Other: Bortezomib
- Cohort 3 (Experimental): AMG 655 (intermediate dose) with Bortezomib
  Interventions: Drug: AMG 655; Other: Bortezomib

INTERVENTIONS:
Drug: AMG 655 — AMG 655 is an investigational, fully human monoclonal agonist antibidy that selectively binds to Death Receptor-5 (DR-5).
Other: Vorinostat — Vorinostat, a second generation polarplanar compound, binds to the catalytic domain of the histone deacetylases (HDAC).
  Other Names: SAHA
  Arms: Cohort 2; Cohort 4; Cohort 6
Other: Bortezomib — A dipeptide boronic acid analogue with antineoplastic activity.
  Other Names: Velcade
  Arms: Cohort 1; Cohort 3; Cohort 5; Cohort 7

SUMMARY:
This is a multi-center, phase 1b study of AMG 655 in combination with bortezomib or vorinostat in subjects with relapsed or refractory low grade lymphoma, mantle cell lymphoma, diffuse large cell lymphoma, and Hodgkin's disease.

Part 1 is an open-label, dose-escalation phase (3+3 design) to determine the safety, tolerability and maximum tolerated dose of AMG 655 in combination with bortezomib or vorinostat. Subjects will be enrolled into one of two arms based on investigator selection (either the bortezomib + AMG 655 arm or vorinostat + AMG 655 arm).

Part 2 of the study is a dose expansion phase that will commence after dose selection of AMG 655 in combination with bortezomib in Part 1. In Part 2, subjects (n = 20) with mantle cell lymphoma will be given AMG 655 in combination with bortezomib. The dose of AMG 655 used in combination with bortezomib will be based on safety and pharmacokinetic information obtained from Part 1 as well as from ongoing AMG 655 trials.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Subjects must have a pathologically confirmed diagnosis of lymphoma that is relapsed or refractory to standard treatment or for which no curative therapy is available. Lymphoma subtypes that are eligible for enrollment include low grade lymphoma, mantle cell lymphoma, diffuse large cell lymphoma, and Hodgkin's disease.
* Part 2: Subjects must have relapsed or refractory mantle cell lymphoma with at least one objective measurable disease site (ie, measurable in at least 2 perpendicular parameters). Subjects must have had at least one prior antineoplastic therapy, up to a maximum of 3. At least one therapy must have included an anthracycline. Subjects must have had documented relapse or progression following the last therapy (ie, most recent therapy given prior to enrollment). An abnormal PET scan will not constitute evaluable disease, unless verified by CT or MRI scan).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic, renal, hepatic and coagulation function

Exclusion Criteria:

* A history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years.
* A history of allogeneic stem-cell transplantation
* Primary central nervous system (CNS) tumors including primary CNS lymphoma
* Central nervous system involvement by lymphoma
* Myocardial infarction within 6 months before enrollment, symptomatic congestive heart failure (New York Heart Association >class II), unstable angina, or unstable cardiac arrhythmia requiring medication
* Vorinostat cohorts only: History of significant GI surgery or disease, which would impair intestinal absorption
* Vorinostat cohorts only: Active peptic ulcer disease
* Prior exposure to AMG 655 or other investigational TRAIL receptor agonists is not permitted
* Prior treatment with bortezomib or vorinostat is not permitted for subjects enrolling in the bortezomib and vorinostat cohorts, respectively
* Major surgery within 28 days before the first dose of AMG 655

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-02; Primary Completion 2010-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Part 1: Safety: Subject incidence of treatment emergent adverse events, Dose Limiting Toxicities, the severity of adverse events and clinically significant changes in safety laboratory tests, physical examinations, or vital signs. | Length of Study
Part 2: Objective response rate of AMG 655 Therapy as determined by using IWG criteria at the dose selected in Part 1, in combination with Bortezomib in subjects with mantle cell lymphoma | Length of Study

SECONDARY OUTCOMES:
Part 2: Overall survival (OS). | Length of study.
Part 2: Progression-Free Survival (PFS). | Length of treatment phase.
Part 2: PK parameters for AMG 655 on a 3 week dosing schedule. | Treatment and follow up phase of study.
Part 2: Subject incidence of anti-AMG 655 antibody formation. | Treatment and follow up phase of study.
Part 2: Duration of response. | Length of treatment phase.
Part 1: Subject incidence of anti-AMG 655 antibody formation. | Treatment and follow up phase of study.
Part 1: Best tumor response, objective response rate and duration of response. | Length of treatment phase.
Part 1: Maximum tolerated dose of AMG 655 administered with bortezomib or vorinostat, if reached. | First 21 days of treatment for each cohort.
Part 1: PK parameters for AMG 655 on a 3 week dosing schedule. | Treatment and follow up phase of study.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Younes A, Sokol L, Ribeiro de Oliveira M, Popplewell L, Romaguera JE, Copeland A, Sabin T, Hsu CP, Pan Y, Gorski K, Hwang Y, Wong S, Beaupre D, Kirschbaum MH.A Phase 1b Study Simultaneously Evaluating Two Novel Conatumumab-Based Combinations in Patients With Relapsed or Refractory Lymphoma.Journal-001239;
- [Background] Younes A, Sokol L, Ribeiro de Oliveira M, Popplewell L, Romaguera JE, Copeland A, Sabin T, Hsu CP, Pan Y, Gorski K, Hwang Y, Wong S, Beaupre D, Kirschbaum MH.A Phase 1b Study Simultaneously Evaluating Two Novel Conatumumab-Based Combinations in Patients With Relapsed or Refractory Lymphoma.Journal-004521;
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com